CLINICAL TRIAL: NCT03828760
Title: Tuning Out: The Effectiveness of Music on Pain and Anxiety in Intrauterine Device Insertion
Brief Title: The Effectiveness of Music on Pain and Anxiety in IUD Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Robin Lennox, Assistant Professor and Family Physician, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Tuning Out
Record Dates: First submitted 2019-01-03; First posted 2019-02-04 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: IUD Insertion Complication; Pain, Acute; Anxiety Acute
Keywords: Intrauterine Device; IUD; Anxiety; Pain; Music; Contraception; Visual analog scale; VAS
MeSH Terms: conditions — Acute Pain; Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and statisticians performing final data analysis will be blinded to the group allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Listening (Experimental): Patients will receive music of choice to listen to using a music-playing device in the waiting room prior to IUD insertion, as well as during the procedure.
  Interventions: Behavioral: Music listening
- Standard Care (No Intervention): Patients will receive standard care (excluding the use of music) from providers at the clinic to minimize pain and anxiety during the procedure.

INTERVENTIONS:
Behavioral: Music listening — Patients will be asked to either use their personal phones to listen to preferred music which is already on their device, or if they do not have a phone or other personal device capable of playing music of their choice, we will use a device (e.g. iPod) to load music of their choice. While in the waiting room, participants will listen to music through headphones/earphones, however they will need to remove their headphones/earphones during the initial consultation with the family physician (explaining risks, etc.), and resume listening to music through the phone speakers once in the examination room as patients will need to be able to hear instructions from the physician during the procedure.
  Arms: Music Listening

SUMMARY:
Although intrauterine devices (IUDs) are a highly effective contraceptive method, fear of pain during insertion is one barrier to use. A review of literature reveals little investigation of interventions for anxiety management during the procedure. Furthermore, evidence of non-pharmacological interventions for both anxiety and pain management is limited. Music has been shown to be effective at reducing anxiety and pain in a variety of contexts, however to the investigators' knowledge, its effectiveness for anxiety and pain relief during the IUD insertion procedure has not been formally examined. This study will therefore examine the effectiveness of listening to music on anxiety and pain during IUD insertion.

DETAILED DESCRIPTION:
The study is a randomized controlled trial of patients at least 16 years of age undergoing an IUD insertion. The experimental group will receive music, self-selected, with a music-playing device prior and during the procedure and the control group will receive standard care. Data for pain and anxiety will be collected prior to the procedure, and during, and after IUD insertion. In addition, a post-procedure questionnaire will be given to patients and providers to ask about satisfaction and acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of English to complete questionnaires
* Women who will attend the clinic for an IUD insertion and accept to participate in the study

Exclusion Criteria:

* Women with chronic pain

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported anxiety (in the moment) | Baseline, immediately after the procedure, immediately after uterine sounding
  100 mm visual analog scale (VAS) measures anxiety reported by patients; values range 0-100 with higher values representing higher anxiety.

SECONDARY OUTCOMES:
Change in self-reported pain (in the moment) | Baseline, immediately after uterine sounding, immediately after insertion, immediately after the procedure
  100 mm visual analog scale (VAS) measures pain reported by patients; values range 0-100 with higher values representing higher pain.
Change in anxiety | Baseline, immediately after the procedure
  The trait anxiety subscale of the State-Trait Anxiety Inventory (Spielberger et al.,1983) will be used to measure trait anxiety. It contains 20 items, each item is rated on a 4-point scale (not at all, somewhat, moderately so, very much so), with higher values representing higher anxiety. Scores range from 20-80 (higher scores represent higher trait anxiety).
Complications related to IUD insertion procedure | Immediately after the procedure
  Patients and providers are asked to identify any significant adverse reactions experienced (by the patient) during the IUD insertion procedure (e.g., bleeding, vasovagal responses) with open-ended survey developed for the study.

OTHER OUTCOMES:
Perceived facilitators and barriers | At study end, approximately 4 months
  Open-ended questionnaire developed for the study asking the provider whether there are any methods to help implement listening to music during the IUD insertion procedure.
Provider satisfaction and acceptability | At study end, approximately 4 months
  Open-ended questionnaire developed for the study asking provider about their opinions regarding the use of music during IUD insertion, whether they would recommend the intervention to patients.
Patient satisfaction and acceptability | Immediately after the procedure
  Open-ended questionnaire developed for the study asking patient about their opinions regarding the use of music during IUD insertion, whether they would recommend the intervention to friends.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Lennox, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Family Practice, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided